CLINICAL TRIAL: NCT02803008
Title: Sun Protection Factor (SPF) Assay: UVA Protection Factor Assay (UVAPF), Minimal Persistent Pigment-Darkening Dose (MPPD)
Brief Title: Sun Protection Factor Assay
Acronym: SPF Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18629
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY987517 (Experimental): Each test site area is divided into test subsite areas that are approximately at least 0.5 cm*2. The application of test material is 2 mg/cm*2. Thus, each 50 cm*2 test site area of a subject requires 100 mg of a test material to obtain a standard 2 mg/cm*2 test application.
  Interventions: Drug: Coppertone (BAY987517)

INTERVENTIONS:
Drug: Coppertone (BAY987517) — Each 50 cm*2 test site area of a subject requires 100 mg of a test material to obtain a standard 2 mg/cm*2 test application. (Formulation number - SR15-46-Z13-072)

SUMMARY:
To evaluate the Sun protection factor efficacy on human skin.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type l, ll and/or lll for UVB testing. Fitzpatrick Skin Type ll, lll and/or lV for UVA testing.
* Male and female
* Aged between 18-70 years old.
* Good health as determined from the HRL SHF(Self History Form)
* Signed and dated Informed Consent Form
* Signed and dated HIPAA (Health Insurance Portability and Accountability Act) Form
* An unbambiguous MED (Minimal Erythema Dose) or MPPD (Minimal Persistent Pigment Darkening Dose)

Exclusion Criteria:

* Subjects on test at any other research laboratory or clinic.
* Known allergy or sensitivity to sunscreens, cosmetics and toiletries, topical drugs and/or ultraviolet light.
* Pre-existing dermatologic conditions which have been diagnosed by a medical professional (e.g. psoriasis, eczema, etc.) which would interfere with this study.
* Pre-existing other medical conditions (e.g. adult asthma. diabetes).
* Treatment with antibiotics within two weeks prior to initiation of the test.
* Chronic medication which could affect the results of the study.
* Known pregnant or nursing women.
* Treatment with antihistamines or corticosteroids within one week prior to initiation of the test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Minimal Erythema Dose (MED) | Up to 15 minutes
Minimal Persistent Pigment Darkening Dose (MPPD) | Up to 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Union, New Jersey, United States